CLINICAL TRIAL: NCT00279383
Title: OSHES (Observational Study on Hemostasis in Surgery ). A Non Interventional Study on the Hemostasis Supportive Methods in Surgery
Brief Title: OSHES - Observational Study on Hemostasis in Surgery (TC-022-IT)
Status: Completed | Type: Observational
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Clinical Trial Operations
Other Study IDs: TC-022-IT
Record Dates: First submitted 2006-01-12; First posted 2006-01-19 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2009-01

CONDITIONS: Blood Loss, Surgical; Hemostasis
Keywords: Intra-operatively treated patients with hemostatic supporting agents/techniques in addition to the standard surgical procedures
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Fibrinogen; Thrombin; TachoSil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fibrinogen (human) + thrombin (human) (TachoSil) — Intra-operatively treated patients with hemostatic supporting agents/techniques in addition to the standard surgical procedures

SUMMARY:
OSHES (= Observational Study on Hemostasis in Surgery) is a non interventional register settled in Italy with the purpose of collecting data on 800 patients intra-operatively treated with hemostatic supporting agents/techniques in addition to the standard surgical procedures in 40 surgical wards. The availability of these data will allow for a better understanding of the therapeutic needs in the area of hemostatic supporting agents/techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are candidates for a specific type of surgery where a supportive hemostyptic agent will be used and who issued an informed consent. A special procedure will be implemented for use in emergency situations.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are candidates for a specific type of surgery where a supportive hemostyptic agent will be used and who issued an informed consent. A special procedure will be implemented for use in emergency situations.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2005-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquarters
Locations (1):
- Nycomed, Roskilde, Denmark